CLINICAL TRIAL: NCT01037192
Title: Evaluating the Use of Large-dose, Extended Interval Vancomycin Intravenous Administration for Skin and Soft Tissue Infections
Acronym: VOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, Anna Yuen, Pharmacist, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VOD
Record Dates: First submitted 2009-12-18; First posted 2009-12-22 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Skin and Soft Tissue Infections
Keywords: outpatient; skin and soft tissue infections; vancomycin intravenous
MeSH Terms: conditions — Soft Tissue Infections | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vanco once daily (Experimental): Subject receives vancomycin 30 mg/kg dose
  Interventions: Drug: vancomycin
- Vanco twice daily (Active Comparator): Subject receives vancomycin 15 mg/kg twice daily
  Interventions: Drug: vancomycin

INTERVENTIONS:
Drug: vancomycin — vancomycin 30 mg/kg intravenous administered once daily
  Arms: Vanco once daily
Drug: vancomycin — vancomycin 15 mg/kg intravenous administered twice daily (standard dosing)
  Arms: Vanco twice daily

SUMMARY:
Our hypothesis is that large-dose, extended-interval vancomycin (30 mg/kg IV q24h) administration provides non-inferior clinical efficacy and microbiological efficacy to standard vancomycin (15 mg/kg IV q12h) administration for skin and soft tissue infections in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 70 years
* Weight 40 - 80 kg
* Suspected or confirmed skin or soft tissue infection for which vancomycin is indicated
* Subject referred to or admitted into OPAT by an Infectious Disease Specialist or Emergency Physician
* Subject able to provide informed consent

Exclusion Criteria:

* Known history of allergy to vancomycin
* Pregnancy
* Granulocytopenia (< 1x109/L)
* Renal impairment (serum creatinine > 177 µmol/L or eGFR < 50 mL/min)
* Known history of vestibular disease or hearing loss
* Subjects treated with vancomycin within the previous month
* Subjects who have received more than 24 hours of vancomycin
* Subjects receiving other antimicrobials that cover MRSA (e.g. cotrimoxazole, rifampin, linezolid)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Yuen, BSc. Pharm, Principal Investigator — Fraser Health
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

REFERENCES:
- [Result] Cohen E, Dadashev A, Drucker M, Samra Z, Rubinstein E, Garty M. Once-daily versus twice-daily intravenous administration of vancomycin for infections in hospitalized patients. J Antimicrob Chemother. 2002 Jan;49(1):155-60. doi: 10.1093/jac/49.1.155. PMID 11751780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from March to September 2010 from patients from the Outpatient Antibiotic Intravenous Therapy clinic at the Royal Columbian Hospital, New Westminster, BC, Canada.
Pre-assignment Details: Subjects were excluded from the trial based on the inclusion and exclusion criteria. The main reasons for exclusion include age and weight.
Groups:
- Vancomycin Once Daily: Subject receives vancomycin 30 mg/kg dose
- Vancomycin Twice Daily: Subject receives vancomycin 15 mg/kg twice daily
Period: Overall Study
Arm/Group | Vancomycin Once Daily | Vancomycin Twice Daily
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vancomycin Once Daily | Vancomycin Twice Daily | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12) | 49 | 48 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Efficacy
Description: Clinical efficacy is determined on the fifth and last day of therapy and is defined favourable if there is resolution of symptoms of infection, return to normal body temperature for at least 48 hours, and normalization or a decrease (> 15%) in leukocytes.
Time Frame: 5 days
Measure: Number; unit: participants
Units Other Than Participants: subjects
Groups:
- Vancomycin Once Daily: Vancomycin 30 mg/kg IV daily
- Vancomycin Twice Daily: Vancomycin 15 mg/kg IV twice daily
Arm/Group | Vancomycin Once Daily | Vancomycin Twice Daily
Number analyzed (Participants) | 3 | 1
Number analyzed (subjects) | 3 | 1
participants | 2 | 0

2. Secondary Outcome: Microbiological Efficacy
Description: Microbiological efficacy is defined as favourable if a repeat culture is negative, if no more materail was obtainable for culture, or if a new microorganism is cultured without clinical signs of infection. It is defined as unfavourable when repeat cultures are positive for the same microorganism, when a new microorganism is cultured with clinical signs of infection or when vancomycin resistance develops. It is defined as indeterminate when the patient is treated with another antibiotic to which the microorganism is susceptible or when no microorganism was cultured at the start of therapy.
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | Vancomycin Once Daily | Vancomycin Twice Daily
Number analyzed (Participants) | 3 | 1
participants
  Favourable | 0 | 0
  Unfavourable | 1 | 0
  Indeterminate | 2 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: March 1 to September 30, 2010
Arm/Group | Vancomycin Once Daily | Vancomycin Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
The main limitation was low enrollment, primarily caused by stringent inclusion criteria. The age limitation was required to ensure safe vancomycin administration. The weight limitation was required for medication preparation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No